CLINICAL TRIAL: NCT00068601
Title: Phase III Trial of LHRH Analog Administration During Chemotherapy to Reduce Ovarian Failure Following Chemotherapy in Early Stage, Hormone-Receptor Negative Breast Cancer
Brief Title: S0230 Goserelin in Preventing Ovarian Failure in Women Receiving Chemotherapy for Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network); Eastern Cooperative Oncology Group (Network); ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000327758; S0230 (Other: SWOG); CALGB-40401 (Other: CALGB); IBCSG-34-05 (Other: IBCSG); U10CA037429 (NIH); NCT00696267 (obsolete NCT alias)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer; Infertility; Menopausal Symptoms
Keywords: infertility; menopausal symptoms; stage II breast cancer; stage IIIA breast cancer; stage IA breast cancer; stage IB breast cancer; estrogen receptor-negative breast cancer; progesterone receptor-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Infertility | interventions — Cyclophosphamide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Chemotherapy (Active Comparator): Patients receive cyclophosphamide-containing chemotherapy alone.
  Interventions: Drug: cyclophosphamide
- Chemotherapy Plus Goserelin (Experimental): Patients receive goserelin subcutaneously once every 4 weeks beginning 1 week before start of cyclophosphamide-containing chemotherapy. Treatment continues until completion of chemotherapy in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclophosphamide; Drug: goserelin acetate

INTERVENTIONS:
Drug: cyclophosphamide — Part of planned chemotherapy regimen
Drug: goserelin acetate — Given subcutaneously
  Arms: Chemotherapy Plus Goserelin

SUMMARY:
RATIONALE: Goserelin blocks hormone production in the ovaries. It is not yet known whether ovarian suppression using goserelin will prevent ovarian failure (early menopause) in women receiving chemotherapy for breast cancer.

PURPOSE: This randomized phase III trial is studying how well giving goserelin together with chemotherapy works compared with chemotherapy alone in preventing early menopause in women with stage I, stage II, or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the rate of premature ovarian failure in women with stage I-IIIA hormone receptor-negative breast cancer treated with chemotherapy with vs without goserelin.

Secondary

* Compare the rate of ovarian dysfunction in patients treated with these regimens.
* Compare ovarian reserve in patients treated with these regimens.
* Describe the pregnancy rates in patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are stratified according to age (under 40 vs 40 to 49) and planned chemotherapy regimen (3- to 4-month/course anthracycline-based vs 6- to 8-month/course anthracycline-based vs 3- to 4-month/course non-anthracycline-based vs 6- to 8-month/course non-anthracycline-based). Patients are randomized to 1 of 2 treatment arms.

* Arm 1: Patients receive cyclophosphamide-containing chemotherapy alone. Patients are followed at 1, 2, and 5 years.
* Arm 2: Patients receive goserelin subcutaneously once every 4 weeks beginning 1 week before start of cyclophosphamide-containing chemotherapy. Treatment continues until completion of chemotherapy in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 416 patients (208 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * Stage I-IIIA
  * Operable disease
* Bilateral synchronous invasive breast cancer allowed provided primary tumors were diagnosed no more than 1 month apart and both tumors are hormone receptor negative
* Must be planning to receive 3-8 months of a preoperative or postoperative chemotherapy regimen containing alkylating agents (anthracyclines or non-anthracyclines), meeting 1 of the following criteria:

  * 3-month/4-course anthracycline-based regimen
  * 6- to 8-month/course anthracycline-based regimen
  * 6- to 8-month/course non-anthracycline-based regimen
* Hormone receptor status:

  * Estrogen receptor negative
  * Progesterone receptor negative

PATIENT CHARACTERISTICS:

Age

* 18 to 49

Sex

* Female

Menopausal status

* Premenopausal

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Fertile patients must use effective barrier contraception
* No other prior malignancy except adequately treated basal cell or squamous cell skin cancer or any in situ cancer from which the patient has been disease-free for at least 5 years after treatment with curative intent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior cytotoxic chemotherapy

Endocrine therapy

* No other concurrent hormonal therapy

Radiotherapy

* Concurrent radiotherapy to the breast, chest wall, or lymph nodes allowed

Surgery

* See Disease Characteristics

Other

* Concurrent participation in other therapeutic clinical trials, including SWOG-S0221, allowed

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 257 (Actual)
Dates: Start 2003-10; Primary Completion 2014-01 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Halle C Moore, MD, Principal Investigator — The Cleveland Clinic; Kathy S. Albain, MD, Study Chair — Loyola University; Silvana Martino, DO, Study Chair — Saint John's Cancer Institute; Ann H. Partridge, MD, MPH, Study Chair — Dana-Farber Cancer Institute; Lori J. Goldstein, MD, Study Chair — Fox Chase Cancer Center; Kelly-Anne Phillips, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (34):
- Australia (14):
  - Mater Hospital - North Sydney, North Sydney, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Newcastle Mater Misericordiae Hospital, Waratah, New South Wales
  - Royal Adelaide Hospital Cancer Centre, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Ballarat Oncology and Haematology Services, Ballarat, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Center - Clayton Campus, Clayton, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Maroondah Hospital, East Ringwood, Victoria
  - St. Vincent's Hospital - Melbourne, Fitzroy, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Belgium (6):
  - Centre Hospitalier Hutois, Huy
  - U.Z. Gasthuisberg, Leuven
  - Centre Hospitalier Regional de la Citadelle, Liège
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
  - AZ Damiaan, Ostend
  - Centre Hospitalier Peltzer-La Tourelle, Verviers
- National Institute of Oncology, Budapest, Hungary
- Italy (5):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Ospedale degli Infermi - ASL 12, Biella
  - Ospedale Civile Ramazzini, Carpi
  - Ospedale Alessandro Manzoni, Lecco
  - European Institute of Oncology, Milan
- Auckland City Hospital, Auckland, New Zealand
- Switzerland (7):
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Inselspital Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Oncology Institute of Southern Switzerland - Locarno, Locarno
  - Oncology Institute of Southern Switzerland - Lugano, Lugano
  - Oncology Institute of Southern Switzerland - Mendrisio, Mendrisio
  - Regionalspital, Thun

REFERENCES:
- [Derived] Moore HC, Unger JM, Phillips KA, Boyle F, Hitre E, Porter D, Francis PA, Goldstein LJ, Gomez HL, Vallejos CS, Partridge AH, Dakhil SR, Garcia AA, Gralow J, Lombard JM, Forbes JF, Martino S, Barlow WE, Fabian CJ, Minasian L, Meyskens FL Jr, Gelber RD, Hortobagyi GN, Albain KS; POEMS/S0230 Investigators. Goserelin for ovarian protection during breast-cancer adjuvant chemotherapy. N Engl J Med. 2015 Mar 5;372(10):923-32. doi: 10.1056/NEJMoa1413204. PMID 25738668
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Chemotherapy | Chemotherapy Plus Goserelin
Started | 131 | 126
Completed | 69 | 66
Not Completed | 62 | 60
Not completed — Ineligible | 11 | 13
Not completed — Not evaluable: withdrew consent | 5 | 4
Not completed — Not evaluable: hysterectomy/oophorectomy | 2 | 4
Not completed — Death | 11 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Missing primary outcome data | 30 | 34

BASELINE CHARACTERISTICS:
Population: Patients who are both eligible and evaluable
Groups:
- Arm 1: Patients receive cyclophosphamide-containing chemotherapy alone.
  cyclophosphamide: Part of planned chemotherapy regimen
- Arm 2: Patients receive goserelin subcutaneously once every 4 weeks beginning 1 week before start of cyclophosphamide-containing chemotherapy. Treatment continues until completion of chemotherapy in the absence of disease progression or unacceptable toxicity.
  cyclophosphamide: Part of planned chemotherapy regimen
  goserelin acetate: Given subcutaneously
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 113 | 105 | 218
Age, Continuous [Median (Full Range); unit: years] | 38.7 [25.1 to 49.9] | 37.6 [26.1 to 48.6] | 37.7 [25.1 to 49.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 105 | 218
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Premature Ovarian Failure at 2 Years
Description: Ovarian failure at two years is defined as amenorrhea (absence of menstrual bleeding) for the preceding six months AND the presence of follicle-stimulating hormone (FSH) in the post-menopausal range.
Time Frame: 2 years
Population: Patients who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Chemotherapy | Chemotherapy Plus Goserelin
Number analyzed (Participants) | 69 | 66
Participants | 15 | 5

2. Secondary Outcome: Rate of Ovarian Dysfunction at 2 Years
Description: Ovarian dysfunction is defined as amenorrhea for the preceding three months and the presence of FSH, estradiol and/or inhibin B levels in the postmenopausal range.
Time Frame: 2 years
Population: Patients with both menstrual status data and at least two available laboratory values (FSH, inhibin B, or estradiol levels) at year 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Chemotherapy | Chemotherapy Plus Goserelin
Number analyzed (Participants) | 67 | 63
Participants | 22 | 9

3. Other Pre Specified Outcome: Ovarian Reserve at 1 and 2 Years
Description: Measurements of ovarian reserve will consist of "Day 2 - 4" levels of FSH, estradiol and inhibin B during Month 12/13 and Month 24/25 (or if amenorrheic, anytime during Month 12/13 and Month 24/25).
Time Frame: 1 and 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Rate of Ovarian Dysfunction at 1 Year
Description: as for outcome 2
Time Frame: 1 year
Population: Patients with both menstrual status data and at least two available laboratory values (FSH, inhibin B, or estradiol levels) at year 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Chemotherapy | Chemotherapy Plus Goserelin
Number analyzed (Participants) | 75 | 78
Participants | 28 | 18

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: This analysis includes all eligible patients who were evaluated for adverse events.
Groups:
- Standard Chemotherapy: Patients receive cyclophosphamide-containing chemotherapy alone. cyclophosphamide: Part of planned chemotherapy regimen
- Chemotherapy Plus Goserelin: Patients receive goserelin subcutaneously once every 4 weeks beginning 1 week before start of cyclophosphamide-containing chemotherapy. Treatment continues until completion of chemotherapy in the absence of disease progression or unacceptable toxicity. cyclophosphamide: Part of planned chemotherapy regimen. goserelin acetate: Given subcutaneously
Arm/Group | Standard Chemotherapy | Chemotherapy Plus Goserelin
Serious Adverse Events (participants affected / at risk) | 0/111 | 1/103
Other Adverse Events (participants affected / at risk) | 70/111 | 73/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Chemotherapy (N=111) | Chemotherapy Plus Goserelin (N=103)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Chemotherapy (N=111) | Chemotherapy Plus Goserelin (N=103)
Nausea (Gastrointestinal disorders) | 9 | 5
Fatigue (asthenia, lethargy, malaise) (General disorders) | 10 | 8
Osteoporosis (Musculoskeletal and connective tissue disorders) | 9 | 1
Pain - Head/headache (Nervous system disorders) | 36 | 36
Libido (Psychiatric disorders) | 27 | 22
Mood alteration - agitation (Psychiatric disorders) | 26 | 19
Mood alteration - anxiety (Psychiatric disorders) | 27 | 31
Mood alteration - depression (Psychiatric disorders) | 36 | 28
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 3 | 12
Vaginal dryness (Reproductive system and breast disorders) | 26 | 30
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 31 | 34
Hot flashes/flushes (Vascular disorders) | 48 | 62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less